CLINICAL TRIAL: NCT03704948
Title: Promoting Emotional Well-Being in Distressed NICU (Neonatal Intensive Care Unit) Mothers: A Phase 2 Evaluation of a Nurse-Delivered Approach
Brief Title: Listening Visits for Emotionally Distressed Mothers of Hospitalized Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201805961; R21NR016751 (NIH)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Nurse Delivered Counseling; Emotional Distress
Keywords: Depression; Listening Visits; Nurses; Hospitalized newborns
MeSH Terms: conditions — Depression | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: We enrolled 55 participants. For the first 45, the study model was parallel. Group 1 received Listening Visits and Group 2 received usual mental health care from a NICU social worker. After study modification design due to the pandemic, the study model was changed to singe group and they received Listening Visits over zoom from a NICU nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial #1: (RCT) Treatment Group: Listening Visits delivered by NICU nurse in person (Experimental): Listening Visits delivered by a NICU nurse in person in the RCT
  Interventions: Behavioral: RCT Treatment -Listening Visits delivered by NICU nurse in person
- Trial #1: (RCT): Control Group -Mental health care delivered by NICU social work (Active Comparator): Mental health care provided by NICU social workers.
  Interventions: Behavioral: RCT Control Usual mental health care delivered by NICU social workers
- Trial #2Open Trial: Listening Visits delivered by NICU nurse over zoom (Experimental): Open Trial: Listening Visits delivered by NICU nurse over zoom
  Interventions: Behavioral: Open trial: Listening Visits delivered by a NICU nurse via zoom

INTERVENTIONS:
Behavioral: RCT Treatment -Listening Visits delivered by NICU nurse in person — 6 sessions, approximately one hour in length, delivered by a nurse who uses empathic listening and problem solving.
  Other Names: Person-centered counselling; Counselling
  Arms: Trial #1: (RCT) Treatment Group: Listening Visits delivered by NICU nurse in person
Behavioral: RCT Control Usual mental health care delivered by NICU social workers — RCT Control Usual mental health care delivered by NICU social workers
  Other Names: Usual Mental Health Care
  Arms: Trial #1: (RCT): Control Group -Mental health care delivered by NICU social work
Behavioral: Open trial: Listening Visits delivered by a NICU nurse via zoom — Open trial: Listening Visits delivered by a NICU nurse via zoom
  Other Names: Person-centered counselling
  Arms: Trial #2Open Trial: Listening Visits delivered by NICU nurse over zoom

SUMMARY:
The proposed research has potential to dramatically improve care for emotionally distressed mothers of newborns hospitalized on the neonatal intensive care unit (NICU). Clinical NICU nurses are well-positioned to provide emotional support in the form of Listening Visits. Specifically, these nurses are easily accessible to NICU mothers, are often the most trusted professional on the healthcare team, they are knowledgeable about the newborn's medical conditions, and, finally they are already skilled in the art of warm communication. This intervention should not only improve depressive outcomes in emotionally distressed NICU mothers but also indirectly impact maternal perception of nurse support which is in turn related to depression symptoms and patient satisfaction, as well as infant length of stay by accelerating maternal readiness for infant discharge.

DETAILED DESCRIPTION:
Infant admission to the neonatal intensive care unit (NICU) is an extremely stressful postpartum outcome, as evidenced by data showing significant depressive symptoms in some 63% of new NICU mothers. Thus, as part of a Family-Centered Care philosophy, focus on the emotional well-being of the mother (and indeed the entire family) should be widely adopted by NICU nursing units. In current clinical practice, however, the emotional well-being of NICU mothers is often ignored. At best, NICU mothers are screened for depression and if indicated, referred to a mental health professional. The extremes of no treatment and full-on mental healthcare comprise an inadequate approach for treating mothers dealing with a normative reaction to a stressful event. In alignment with the Nurse Parent Support Model, the investigators propose the implementation of Listening Visits as a cost-effective nurse-delivered supportive approach, proven to relieve moderately severe depressive symptoms in mothers of term infants. In the NICU setting, Listening Visits were first implemented in a phase-1 feasibility trial conducted by this research team. In that first trial, Listening Visits were delivered by a doctoral-level nurse practitioner and showed promise as means to reduce distress in NICU mothers. A Listening Visit program for emotionally distressed NICU mothers is innovative because it is a cost-effective approach that uses resources that are largely in place, to serve a persistent unmet need in a vulnerable postpartum population. By having nurses provides support, the concept of emotional distress in NICU mothers is normalized. This new application of Listening Visits also directly aligns with the NINR emphasis on promoting coping to prevent compromising mood states. The promising results of the feasibility trial now must be challenged with a control group comparison to definitively attribute maternal improvements to Listening Visits. Thus the objective of the proposed research is to conduct a Phase 2 pilot RCT to evaluate Listening Visits provided by bachelor's-level NICU nurses as compared with the care currently provided by the NICU social work team. The investigators will assess the relative effectiveness of Listening Visits vs. standard care on depressive symptoms. 50 women will be randomized into this trial.Due to the pandemic, recruitment for the RCT was halted with 45 women enrolled. Enrollment to the RCT of Listening Visits is closed.

With approval from NINR, the IRB protocol of the RCT was modified to an open trial design, in which women received Listening Visits from a NICU nurse via Zoom. The goal is to enroll 20 women. In consultation with the Human Subjects Office University of Iowa (who in turn consulted with staff of Clinical Trials.gov), the study design section of this clinical trials registration number is updated to reflect the ongoing open trial design.

We enrolled 55 participants. For the first 45, the study model was parallel. Group 1 received Listening Visits and Group 2 received usual mental health care from a NICU social worker. After the study modification design due to the pandemic, the study model was changed to a single group and they received Listening Visits over Zoom from a NICU nurse. We have listed the three arms based on both study designs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and read English
* 18 years of age or older Edinburgh Postnatal Depression Scale (EPDS) score= 12 through 19, inclusive; with a rating of 2 or less on EPDS item #10)
* Hospitalized newborn

Exclusion Criteria Women is not currently receiving counseling services

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S. Segre, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Stead Family Children's Hospital, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segre LS, Brock RL, O'Hara MW. Depression treatment for impoverished mothers by point-of-care providers: A randomized controlled trial. J Consult Clin Psychol. 2015 Apr;83(2):314-24. doi: 10.1037/a0038495. Epub 2014 Dec 8. PMID 25486371
- [Background] Segre LS, Chuffo-Siewert R, Brock RL, O'Hara MW. Emotional distress in mothers of preterm hospitalized infants: a feasibility trial of nurse-delivered treatment. J Perinatol. 2013 Dec;33(12):924-8. doi: 10.1038/jp.2013.93. Epub 2013 Aug 15. PMID 23949835

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events after participant enrollment.
Groups:
- Trial #1 (RCT) Treatment Group: Listening Visits Delivered by NICU Nurse in Person: Listening Visits delivered by a NICU nurse in person in the RCT
  RCT Treatment -Listening Visits delivered by NICU nurse in person: 6 sessions, approximately one hour in length, delivered by a nurse who uses empathic listening and problem solving.
- Trial #1 (RCT) Control Group: Usual Mental Health Care Delivered by NICU Social Work: Mental health care provided by NICU social workers.
  RCT Control Usual mental health care delivered by NICU social workers: RCT Control Usual mental health care delivered by NICU social workers
- Trial #2 (Exploratory Open Trial Due to Pandemic) Listening Visits Delivered Via Zoom: Open trial of Listening Visits delivered by NICU nurses via zoom. When Trial 1 (RCT) was halted because of the pandemic, we conducted a small, open trial evaluating Listening Visits delivered by NICU nurses via zoom.
Period: Overall Study
Arm/Group | Trial #1 (RCT) Treatment Group: Listening Visits Delivered by NICU Nurse in Person | Trial #1 (RCT) Control Group: Usual Mental Health Care Delivered by NICU Social Work | Trial #2 (Exploratory Open Trial Due to Pandemic) Listening Visits Delivered Via Zoom
Started | 22 | 23 | 10
Completed | 20 | 22 | 9
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Trial #1 (RCT) Control Group: Mental Health Care Delivered by NICU Social Work: Mental health care provided by NICU social workers.
  RCT Control Usual mental health care delivered by NICU social workers: RCT Control Usual mental health care delivered by NICU social workers
- Trial #2 (Open Trial Due to Pandemic) Listening Visits Delivered Via Zoom by a NICU Nurse: Trial 1, the RCT (Arms 1 and 2) were halted because of the pandemic with 45 of the 50 projected participants enrolled. We closed enrollment to the RCT and pivoted (with NINR approval) conduct an exploratory open trial of Listening Visits delivered via zoom by a NICU nurse.
  As directed by NIH help desk, the data for Arm 3 (the open trial of Listening Visits delivered via zoom by a NICU nurse) is reported here as "Arm 3."
- Total: Total of all reporting groups
Arm/Group | Trial #1 (RCT) Treatment Group: Listening Visits Delivered by NICU Nurse in Person | Trial #1 (RCT) Control Group: Mental Health Care Delivered by NICU Social Work | Trial #2 (Open Trial Due to Pandemic) Listening Visits Delivered Via Zoom by a NICU Nurse | Total
Number analyzed (Participants) | 20 | 22 | 9 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 9 | 51
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 9 | 51
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 22 | 9 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 17 | 16 | 7 | 40
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 22 | 9 | 51
Mean Score IDAS-GD [Mean (Standard Deviation); unit: units on a scale] | 53.50 (11.35) | 53.00 (14.12) | 56.89 (11.85) | 53.88 (12.53)

OUTCOME MEASURES:

1. Primary Outcome: Mean IDAS-GD Score at 4 Weeks (End of Treatment) and 8 Weeks (Follow up)
Description: * Scale: Inventory of Depression & Anxiety Symptoms-General Depression (sub) Scale (IDAS-GD).
  * The IDAS-GD assesses depression symptoms
  * The IDAS-GD is a 20-item Likert-scale instrument assesses dysphoria, suicidality, lassitude, insomnia, appetite loss and well-being, using a 5-point scale ranging from not at all to extremely, indicating how much they had experienced each symptom during the past 2 weeks.
  * Total score for IDAS-GD can range from 1-100, with higher scores indicating more depression symptoms
Time Frame: 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trial #1: (RCT) Treatment Group: Listening Visits Delivered by NICU Nurse in Person | Trial #1: (RCT): Control Group -Mental Health Care Delivered by NICU Social Work | Trial #2Open Trial: Listening Visits Delivered by NICU Nurse Over Zoom
Number analyzed (Participants) | 16 | 21 | 9
score on a scale
  4 Weeks (end of treatment) | 46.12 (12.74) | 51.10 (13.32) | 40.11 (13.78)
  8 Weeks (follow up) | 42.39 (12.37) | 41.69 (13.32) | 32.39 (10.04)
Statistical Analysis 1: Comparison: Trial #1: (RCT) Treatment Group: Listening Visits Delivered by NICU Nurse in Person vs Trial #1: (RCT): Control Group -Mental Health Care Delivered by NICU Social Work; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 0.82

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Groups:
- Trial #1 RCT Treatment Group Listening Visits Delivered by NICU Nurses in Person: Trial #1 RCT Treatment Group Listening Visits delivered by NICU nurses in person
- Trial #1 RCT Control Group-Usual Mental Health Care From Social Work: Trial #1 RCT Control Group-Usual mental health care from social work
- Trial #2: Listening Visits Delivered Via Zoom: Trial #2: Listening Visits delivered via zoom
Arm/Group | Trial #1 RCT Treatment Group Listening Visits Delivered by NICU Nurses in Person | Trial #1 RCT Control Group-Usual Mental Health Care From Social Work | Trial #2: Listening Visits Delivered Via Zoom
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/9
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/9

LIMITATIONS AND CAVEATS:
Trial #1: RCT-Small sample, lack of ethnic/racial diversity in the sample, types of treatment used by usual care group was not documented Trial #2: Open Trial: Small, sample, lack of ethnic/racial diversity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03704948/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT03704948/SAP_001.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03704948/ICF_002.pdf